CLINICAL TRIAL: NCT04679532
Title: NBA G-League Sweat Testing Study: Validity of the Gx Sweat Patch in Measuring Sweating Rate and Sweat Chloride Concentration During On-court Training With Basketball Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PepsiCo Global R&D (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PEP-2001
Record Dates: First submitted 2020-12-09; First posted 2020-12-22 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Sweat Analysis
Keywords: sweating rate; sweat electrolytes; sweat electrolyte concentration; sweat patch; wearable; epidermal; Gx patch

STUDY DESIGN:
Intervention Model Description: Each subject serves as their own control. Both devices are worn during the same exercise session.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Validation. Gx sweat collection patch (Other): Left ventral forearm placement using Epicore Biosystems Gx patch
  Interventions: Other: Gx sweat patch
- Validation. Reference sweat collection patch (Other): Right ventral forearm placement using a well-established methodology as published in peer-reviewed journals
  Interventions: Other: Reference sweat patch

INTERVENTIONS:
Other: Gx sweat patch — Adhesive-backed flexible epidermal wearable regional sweat patch to collect and analyze sweat via microfluidics and colorimetric assay
  Arms: Validation. Gx sweat collection patch
Other: Reference sweat patch — Adhesive Tegaderm with absorbent pad regional sweat patch to collect sweat, followed by standard benchtop gravimetry and ion chromatography methods to analyze sweat
  Arms: Validation. Reference sweat collection patch

SUMMARY:
To determine the validity of the Gx Sweat Patch in measuring sweating rate and sweat chloride concentration during moderate-high intensity practice against well-established reference methods in field conditions with basketball athletes

ELIGIBILITY:
Inclusion Criteria:

* 18-40 years of age
* Subject is participating in training/competition with the NBA G-league
* Subject is participating in a coach led practice

Exclusion Criteria:

* Subject has an allergy to adhesives (e.g., experiences rash reactions to typical adhesive bandages)
* Subject has participated in a clinical trial within past 30 days
* Subject has participated in any PepsiCo trial within past 6 months
* Subject has a condition the investigator believes would interfere with his/her ability to provide informed consent, comply with the study protocol, which might confound the interpretation of the study results or put the person at undue risk

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — No females in NBA G-League
Enrollment: 65 (Actual)
Dates: Start 2020-12-08 (Actual); Primary Completion 2021-11-04 (Actual); Study Completion 2021-11-04 (Actual)

PRIMARY OUTCOMES:
Regional sweat chloride concentration | Average across a single practice session on 1 day
  Gx patch vs. reference patch during exercise. Gx patch analyzed by colorimetry via smartphone app. Reference patch analyzed with ion chromatography

SECONDARY OUTCOMES:
Regional sweating rate | Average across the same single practice session on the same 1 day as the primary outcome
  Gx patch vs. reference patch during exercise. Gx patch analyzed by microfluidic reading with Smartphone. Reference patch analyzed with gravimetry
Whole body sweating rate | Measured one time to represent the average across the same single practice session on the same 1 day as the primary outcome
  Change in body mass from pre- to post-exercise, corrected for fluid/food intake and urine loss. Body mass measured to the nearest 0.01 kg using a digital platform scale

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay B Baker, PhD, Principal Investigator — PepsiCo Global R&D, Gatorade Sports Science Institute (GSSI) Barrington, IL
Locations (1):
- NBA G League Ignite Team Site Ultimate Fieldhouse, 2675 Mitchell Dr., Walnut Creek, California, United States

IPD SHARING:
Plan to Share IPD: No